CLINICAL TRIAL: NCT02090647
Title: Aesthetic Outcome of Osseospeed Implants With Three Different Abutment Materials. A Randomized Controlled Clinical Study
Brief Title: Aesthetic Evaluation of Different Abutment Materials for OsseoSpeed Implants
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Siena (Other)
Responsible Party: Principal Investigator, Prof. Marco Ferrari, Professor, University of Siena
Allocation: Randomized | Model: Factorial | Masking: Single | Purpose: Treatment
Other Study IDs: ABTM001
Record Dates: First submitted 2014-03-14; First posted 2014-03-18 (Estimated); Last update posted 2014-03-18 (Estimated); Status verified 2014-03

CONDITIONS: Aesthetic Evaluation; Implant Survival Rate
Keywords: dental implant, aesthetic, implant abutment

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: No

ARMS (5):
- titanium 1 (Active Comparator): titanium abutment type 1
  Interventions: Behavioral: aesthetic outcome
- titanium 2 (Active Comparator): titanium abutment type 2
  Interventions: Behavioral: aesthetic outcome
- zirconia 1 (Active Comparator): zirconia abutment type 1
  Interventions: Behavioral: aesthetic outcome
- zirconia 2 (Active Comparator): zirconia abutment type 2
  Interventions: Behavioral: aesthetic outcome
- titanium nitrate (Active Comparator): titanium nitrate abutment
  Interventions: Behavioral: aesthetic outcome

INTERVENTIONS:
Behavioral: aesthetic outcome

SUMMARY:
The objective of the study was to assess the aesthetic outcome of different abutments materials and shapes on dental implants .

A set of parameters, including assessments of the mucosa and periodontal tissue , soft tissue , radiographic evaluations and clinical photographs, was used to obtain a measure of the aesthetic of implant-prosthesis rehabilitations.

ELIGIBILITY:
Inclusion Criteria:

* aged over 18 years
* dental implant rehabilitation requested
* at least 1 tooth missing in areas between 1.5-3.5 and 3.5-4.5
* sufficient bone volume for implant placement ( length 10-15mm; diameter 2.5-4mm, bone quality between class I and III of Lekholm and Zarb).
* informed consensus acceptance

Exclusion Criteria:

* systemic pathologies that represent controindication to implantology
* smoking (more than 10 cigarettes per day)
* severe bruxism
* untreated periodontitis

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 90 (Actual)
Dates: Start 2012-01; Primary Completion 2013-07 (Actual); Study Completion 2014-01 (Actual)

PRIMARY OUTCOMES:
aesthetic evaluation | 12 months
  measure of how the implant-prosthesis restoration is able to comply with the color, shape and proportions imitating as much as possible natural dentition.

SECONDARY OUTCOMES:
implant survival rate | 12 months
  Survival rate means the success rate of the dental implant and/or the restoration that is placed on top of the dental implant.

CONTACTS AND LOCATIONS:
Locations (1):
- Department of Dental Materials and Fixed Prosthodontics of the University of Siena, Policlinico Le Scotte, Siena, Siena, Italy